CLINICAL TRIAL: NCT03508531
Title: Evaluation of Postoperative Analgesic Effect of Ultrasound Guided Erector Spinae Plane Block and Oblique Subcostal Transverse Abdominis Plane Block in Laparoscopic Cholecystectomy, Randomised Controlled Study
Brief Title: Erector Spinae Plane Block and Oblique Subcostal Transverse Abdominis Plane Block in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Asst. Prof. Serkan Tulgar, M.D., Assistant proffessor, Maltepe University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ESPvsOSTAP
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Controlled randomized study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESP Block (Active Comparator): Ultrasound-guided bilateral Erector spinae plane block performed at end of the surgery with 40 ml of a bupivacaine/lidocaine mixture. Perioperative and postoperative routine analgesic protocol will be performed (consist of intravenous analgesics and intravenous patient-controlled analgesia) with no additional intervention (block) Standard Pain Followup and Monitorization will be performed.
  Interventions: Procedure: ESP Block; Other: Standard Pain Followup and Monitorization
- OSTAP Block (Active Comparator): Ultrasound-guided bilateral OSTAP block performed at end of the surgery with 40 ml of a bupivacaine/lidocaine mixture. Perioperative and postoperative routine analgesic protocol will be performed (consist of intravenous analgesics and intravenous patient-controlled analgesia) with no additional intervention (block) Standard Pain Followup and Monitorization will be performed.
  Interventions: Procedure: OSTAP block; Other: Standard Pain Followup and Monitorization
- Control (Sham Comparator): Perioperative and postoperative routine analgesic protocol will be performed (consist of intravenous analgesics and intravenous patient-controlled analgesia) with no additional intervention (block) Standard Pain Followup and Monitorization will be performed. No block will be performed in this group.
  Interventions: Other: Standard Pain Followup and Monitorization

INTERVENTIONS:
Procedure: ESP Block — A high-frequency linear ultrasound transducer will be placed in a longitudinal parasagittal orientation 3 cm lateral to T9 spinous process. The erector spinae muscles will be identified superficial to the tip of T9 transverse process. The patient's skin will be anesthetized with 2% lidocaine. A 17-gauge 8-cm needle will be inserted using an in-plane superior-to-inferior approach to place the tip into the fascial plane on the deep (anterior) aspect of erector spinae muscle. The location of the needle tip will be confirmed by visible fluid spread lifting erector spinae muscle off the bony shadow of the transverse process. A total of 40 mL of bupivacaine/lidocaine mixture will be injected.
  Arms: ESP Block
Procedure: OSTAP block — The bilateral OSTAP will be performed at the end of the surgery. A total of 40 ml local anesthetic mixture (Bupivacaine and lidocaine) will be injected bilaterally with interfascial plane between the external oblique and transversus abdominis muscles
  Arms: OSTAP Block
Other: Standard Pain Followup and Monitorization — Numeric Rating Scale (NRS) pain score will be recorded from 20th minute in recovery room followed by 1.-3.-6.-12.-18.-24.hours. Intravenous meperidine administration at 0.5 mg / kg rescue analgesia was determined in patients with a NSR score of 6 and over in the postoperative collection room. It is planned that the patient will continue to follow the hourly NRS score in ward. Intramuscular diclofenac will be administered in this period if NRS 6 and if it is over, intravenous 0.5 mg / kg meperidine will be administered if NRS score is 6 or more after 2 hours. Salvage analgesic needs and times will be noted in detail, and the use of rescue analgesics, as well as NRS scores at designated hours, will be kept in a statistical evaluation.

SUMMARY:
Erector Spinae Plane Block is a newly defined regional anesthesia technique. Its use for many indications has been identified by case reports in the literature. As the investigators have considered that erector spinae plane block could be efficacious for providing postoperative analgesia in laparoscopic cholecystectomy, the investigators have implemented the application of this blockade into practice at the clinic.Oblique subcostal transverse abdominis plane block (OSTAP) is another regional anesthesia technic used for postoperative analgesia in laparoscopic cholecystectomy. Main purpose of this study is to compare the analgesic effect of ultrasound-guided erector spinae block and OSTAP in laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

-Elective laparoscopic Cholecystectomy, ASA status 1-2 -

Exclusion Criteria:

* Patient refusal
* Contraindications to regional anesthesia
* Known allergy to local anesthetics
* Bleeding diathesis
* Use of any anti-coagulants
* Inability to provide informed consent
* Severe kidney or liver disease
* Inability to operate PCA system
* Patient with psychiatric disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 Years to 65 Years
Enrollment: 60 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-05-21 (Actual)

PRIMARY OUTCOMES:
Pain | 24 hours
  Changes in Numeric Rating Scale (NRS) at rest and on movement will be recorded at intervals. NRS is a unidimensional measure of pain intensity in adults. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

SECONDARY OUTCOMES:
analgesic consumption | 24 hours
  Tramadol consumption in Patient Controlled Analgesia device and additional and rescue analgesic using

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Tulgar, Ass Prof, Principal Investigator — Maltepe University faculity of medicine
Locations (1):
- Maltepe University faculty of medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aksu C, Gurkan Y. Ultrasound-guided bilateral erector spinae plane block could provide effective postoperative analgesia in laparoscopic cholecystectomy in paediatric patients. Anaesth Crit Care Pain Med. 2019 Feb;38(1):87-88. doi: 10.1016/j.accpm.2018.03.008. Epub 2018 Apr 6. No abstract available. PMID 29630940
- [Background] Basaran B, Basaran A, Kozanhan B, Kasdogan E, Eryilmaz MA, Ozmen S. Analgesia and respiratory function after laparoscopic cholecystectomy in patients receiving ultrasound-guided bilateral oblique subcostal transversus abdominis plane block: a randomized double-blind study. Med Sci Monit. 2015 May 7;21:1304-12. doi: 10.12659/MSM.893593. PMID 25948166